CLINICAL TRIAL: NCT06170905
Title: Effect of Whey Protein on Postprandial Glucose Excursions in Pregnant Women
Brief Title: Whey Protein Pre-load and Postprandial Glycemia in Pregnancy
Acronym: ProGs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Prof. Martin Heni, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 78/23
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Postprandial Glycemia
Keywords: postprandial glucose excursions; glycemia; whey protein; protein pre-load; pregnancy; gestational diabetes mellitus; insulin secretion; incretins
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Each participant will undergo two oral glucose tolerance tests (i) one with whey protein pre-load and (ii) one without, in a randomized order.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral glucose tolerance test with whey protein pre-load (Experimental): 30 minutes prior to the 75 g OGTT, a whey protein solution is given.
  Interventions: Dietary Supplement: Whey protein-preload OGTT
- Control oral glucose tolerance (No Intervention): 75 g OGTT without whey protein pre-load.

INTERVENTIONS:
Dietary Supplement: Whey protein-preload OGTT — Intake of 25 g whey protein diluted in water 30 minutes prior to the start of a regular 75 g oral glucose tolerance test
  Arms: Oral glucose tolerance test with whey protein pre-load

SUMMARY:
This pilot study aims to investigate the intake of whey protein prior to carbohydrate intake as an approach to modulate postprandial glucose excursions during pregnancy.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) has transgenerational health consequences and increases the risk of type 2 diabetes mellitus in both mother and child. However, there is a lack of practical nutritional concepts for the prevention and treatment of GDM. This randomized controlled pilot study investigates whether the intake of a protein drink before carbohydrate intake lowers postprandial blood glucose levels of pregnant women. Therefore, two 75g oral glucose tolerance tests are performed in 20 pregnant women in a cross-over design, whereby a whey protein solution is drunk 30 minutes before one of the oral glucose tolerance tests (OGTT). If a clinically relevant effect on blood glucose levels is identified, this project can clarify whether the reduction in postprandial glycemia was caused by changes in the secretion of insulin and incretins.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24+0 and 27+6 (+/- 7 days) weeks of pregnancy after menstruation
* BMI before pregnancy: 18 - 29.9 kg/m2
* No known underlying diseases
* Understanding and voluntary signing of a consent form before study-related examinations

Exclusion Criteria:

* Age < 18 years
* Diabetes mellitus type 1 or type 2
* Drug therapy that raises or lowers blood sugar, e.g. steroids, antidiabetics, insulin.
* Endocrine disorders (e.g. hyperthyroidism, polycystic ovary syndrome (PCOS), ...)
* Current depression or other mental illnesses
* Eating disorder
* Regular intake of medication other than vitamins/trace elements during pregnancy
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m²
* C-reactive protein > 10 mg/l
* Transaminase elevation of 2 times the upper norm
* Pre-existing cardiac diseases
* Drug and/or alcohol abuse
* Hb < 12 g/dl
* No consent to be informed about incidentally discovered pathological findings
* Any other (clinical) condition that would endanger participants safety or question scientific success according to the physicians opinion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Glucose course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course of plasma glucose assessed during a 75 g oral glucose tolerance test with vs without whey protein pre-load in pregnant women.
Postprandial glucose excursion | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Area under the glucose curve (AUC 0-30 Min. and AUC 0-120 Min.) and peak glucose assessed during a 75 g oral glucose tolerance test with vs without whey protein pre-load in pregnant women.

SECONDARY OUTCOMES:
Insulin course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course of insulin assessed during the 75 g oral glucose tolerance test in pregnant women.
C-peptide course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course C-peptide assessed during the 75 g oral glucose tolerance test in pregnant women.
Insulin secretion | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Insulin secretion assessed during the 75 g oral glucose tolerance test in pregnant women.
Insulin sensitivity | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Insulin sensitivity assessed during the 75 g oral glucose tolerance test in pregnant women.
Glucagon course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course of glucagon and area under the glucagon curve assessed during the 75 g oral glucose tolerance test in pregnant women.
GLP-1 course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course of glucagon-like peptide 1 (GLP-1) and area under the GLP-1 curve assessed during the 75 g oral glucose tolerance test in pregnant women.
GIP course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course of glucose-dependent insulinotropic polypeptide (GIP) and area under the GIP curve assessed during the 75 g oral glucose tolerance test in pregnant women.
Glicentin course | Timepoint 0-120 minutes during the oral glucose tolerance test.
  Course of glicentin and area under the glicentin curve assessed during the 75 g oral glucose tolerance test in pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Martin martin.heni@uniklinik-ulm.de, Prof., Principal Investigator — University Hospital Ulm
Locations (1):
- Universityhospital Ulm, Ulm, Germany